CLINICAL TRIAL: NCT02158962
Title: An Integrated Risk Reduction Intervention for Abused African Caribbean Women
Brief Title: Empowered Sisters Project Making Choices Reducing Risks
Acronym: ESP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Virgin Islands (Other)
Responsible Party: Principal Investigator, Doris W Campbell, PhD, Senior Research Professor, University of the Virgin Islands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: [460913-1]
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Domestic Violence; Domestic Abuse
Keywords: Partner abuse; Abuse African Caribbean women; Intimate Partner Violence
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral - Education (Experimental): 3 Educational Sessions
  Session 1 - Reducing Risk for Intimate Partner Violence (IPV); Session 2 - Reducing risk for Sexually Transmitted Infections including HIV (STI/HIV) Session 3 - A group session which reinforces skills for reducing IPV and STI/ HIV risk reduction.
  Interventions: Behavioral: Behavioral - Education
- Behavioral - Education (Active Comparator): 3 Educational Sessions
  Session 1 - Breast Health Education and Developing A Breast Cancer Risk Reduction Plan Session 2 - Reducing risk for overweight and obesity and Developing a Healthy Eating and Activity Plan Session 3 - A group session which integrates and reinforces skills from Sessions 1 and 2.
  Interventions: Behavioral: Behavioral - Education

INTERVENTIONS:
Behavioral: Behavioral - Education — Behavioral - Education
  3 educational sessions aimed at reducing risks partner violence, and sexual transmitted infections
  Other Names: Education; Skill Building

SUMMARY:
The purpose of this study is to combine a culturally tailored and integrated Risk Reduction Intervention in the US Virgin Islands (USVI) in a clinical trial randomly assigning abused women to a 1) Healthy Relationships experimental group of three sessions of risk reduction interventions or 2) a Healthy Living comparison control group of three session of health promotion activities to determine if the combined, intervention is safe and effective in a test the following hypotheses:

1. Women in the integrated risk reduction intervention will score significantly lower on outcome measures of intimate partner abuse (IPA) and STD/HIV risk behaviors end of Session III and at 3 and 6 months than women in the control group
2. Women in the integrated risk reduction Intervention will score significantly higher on IPA safety behaviors and STI/HIV prevention behaviors at end of Session III and at 3 and 6 months than women in the control group.

Several exploratory and major controlled studies on the mainland US have shown intimate partner violence (IPV) and intimate partner abuse (IPA) to be risk factors for a variety of physical, reproductive and mental health problems, including sexually transmitted infections and HIV/AIDS, many of which are areas of known health disparity for African American and Latina women. A recently completed study of African Caribbean and African American women in the US Virgin Islands revealed that nearly one third of women reported lifetime partner abuse and increased risk for sexually transmitted infections including HIV/AIDS. Abused women in the USVI had significantly more risk factors for HIV/AIDS than did women who were not abused.

The proposed intervention combines an empowerment model designed to help abused women make choices that protect the physical and emotional health of the woman and her family with a sexual safety model designed to help her make choices to reduce her risk of acquiring an STI or contracting HIV/AIDS. The integrated model adapts two interventions that have been tested with African American women on the US mainland and found to be effective as separate interventions for IPV and IPA and reducing the risk of STI/HIV. The adapted interventions will be used with abused African Caribbean women based on an a priori assessment of the cultural attitudes, beliefs and resources available to women living in an island environment with limited resources.

DETAILED DESCRIPTION:
I. Background and Significance: Several exploratory and major controlled studies conducted on the mainland US have shown intimate partner violence (IPV) or intimate partner abuse (IPA) to be risk factors for a variety of physical, reproductive and mental health problems, including HIV/AIDS, many of which are areas of known health disparity for African American and Latina women.

The current investigators recently completed the first in-depth prevalence study of violence and abuse of women in the US Virgin islands (USVI) and associated health consequences. This seminal study showed 1) Lifetime prevalence of IPV of 32.8% in the USVI and past two year prevalence of 37.2%%.in a sample of 1059 women aged 18-55 who self-identified as African Caribbean or from African descent and who had an intimate partner during the past two years 2) Past two year physical and/or sexual abuse ranged from 4 % on the island of St Croix to 9% on St Thomas 3) Abused women had significantly more risk factors for Sexually Transmitted Infections (STIs) and HIV/AIDS than did women not abused, and 4) Risk factors for STIs and HIV/AIDS included being forced into vaginal or anal sex, women having concurrent partners or their partners having multiple partners, having a STI, lack of consistent condom use, and exchange sex (trading sex for material goods) This study also found women amenable to being asked about IPV in health care settings where a brief intervention could be feasibly implemented. Preliminary qualitative work illuminated women's perceptions of community and cultural perspectives on IPV in the USVI. The proposed randomized clinical trial (RCT) builds on findings from the prior study.

II. Research Strategy: A RCT will provide a preliminary test of an intervention designed to reduce IPV and IPA and the concurrent risk of STIs and HIV in abused USVI women by empowering their use of safety behaviors and increasing their use of resources... IPV and IPA have been linked to high-risk sexual behaviors, the inability to negotiate safer sex behaviors, and negative sexual health outcomes. The research plan is to deliver a structured intervention to reduce the devastating impact of IPV and IPA for abused women in the USVI.

Time I: Women will respond to baseline data measures using computer assisted self-reports. Data collected include socio-demographic and cultural characteristics of women and their partners, past and recent intimate partner physical, sexual and emotional abuse (SVAWS), Danger Assessment (DA), baseline HIV/STD status and risks for infection, including condom use. To minimize attrition contact information for each participant and for three contact persons (family, friends, and neighbors) will also be collected. Abused women will be randomized by the computer to either the Healthy Relationships Risk Reduction experimental intervention group or the Healthy Lifestyles comparison control group A. Session 1- Risk Reduction Intervention Group. Women in the Experimental Intervention will complete this session following initial assessment and group assignment. The ESP-DOVE IPV Empowerment Intervention is an individualized (60 minute) protocol following the initial enrollment session. Abused women will view a video developed in the US Virgin Islands, using local actors, depicting various experiences of abused Virgin Island. The abused women will participate in a one on one structured, brochure-based intervention with a trained interventionist that addresses information about the cycle of violence, risk factors that may increase a woman's danger of homicide (the Danger Assessment), choices or options (leaving, using local shelter resources, accessing resources in the criminal justice system), safety planning, and specific local and national phone numbers for IPV resources. The intervention provides the woman with information, emphasizing that she has options or The structured ESP- DOVE intervention is interactive and encourages the woman to describe her experiences and choose her options as they proceed. The intervention has been modified to be culturally appropriate for abused women of African Caribbean or African American background living in the US Virgin Islands. Since the context of IPV varies considerably, this approach allows individualization, client input and choice, all thought to enhance intervention success with battered women and other "hard to reach" populations At the same time, the brochure gives the nurse and other interventionists a script to increase uniformity of the intervention across women and interventionists. Four major intervention components: a) IPV information, b) Danger Assessment, c) Safety Planning, and d) Resources are explored. At the end of Session I, the woman in the risk reduction intervention group will provide contact information for Session 2 which will be scheduled one week later.

Time 2: Session 2- Women will assess their needs associated with IPV, safety behaviors and feelings about how their situation is evolving. The need for resources and services will be explored. The session will also focus on helping the women learn how to reduce their risk for HIV/STD infections. This one-on-one behavioral intervention has been found to reduce HIV/STD risk behaviors and STD morbidity among inner-city African American women in primary care settings in a NINR funded randomized controlled trial. The intervention has been modified and culturally tailored for abused women in the US Virgin Islands and involves a skill-building one-on-one session that the facilitator tailors to the specific needs of each participant after conducting an HIV/STD risk assessment interview. It involves STD prevention behavioral skills, video clips, condom demonstration, practice with an anatomical model, and role-playing. Curriculum activities are also designed to help women recognize that faulty reasoning and decision-making can increase their risk of HIV infection. The activities help the women understand the adverse consequences of participating in unsafe sexual activity and the positive consequences of safer sexual practices. Contact information for Session 3 will be validated and a follow up group session scheduled.

Time 3: Session 3: The third session will consist of small groups (8-10) of women in a supportive/educational session led by an interventionist and investigator. Sessions held in each district in the USVI and will be scheduled two weeks following Session 2. Women in the experimental intervention group will have another opportunity to integrate issues related to their IPV experiences. . They will interact with other abused women in a setting conducive to sharing attitudes and beliefs about IPV prevention, cultural beliefs about IPV, the need for support, assertiveness training, stress and affect management, safety enhancement strategies and effective behaviors to reduce the risk of HIV and sexually transmitted disease and personal vulnerability. Session three will be offered twice each week in each district until all participants have had an opportunity to complete the intervention. At the end of session 3, the women will be scheduled for a three month follow-up to assess outcomes. Contact information will be reconfirmed.

B. Healthy Living Comparison Control Group Session 1: Women in the Healthy Living comparison control group will complete the baseline assessment using the computer assisted tablets for self-report. Women who report a history of intimate partner abuse will be will be yoked on age (>25 or <below 25) and ethnicity (Hispanic or Non-Hispanic and education (HS grad vs < high school graduation). During Session one, if randomly assigned to the Healthy Living Comparison Control intervention group, they will be focus on Breast Health Education and how to develop a breast health care plan aimed at reducing the risk of breast cancer in women of African heritage. Obesity as a risk factor for breast cancer will be introduced. Booklets on breast health and developing a breast health plan will be provided as well as general resource information on women and child health services. Contact information for the one week follow up will be obtained and the woman given an appointment for Session II.

Session 2: At time two women in the comparison control health promotion group will be involved in a session on Healthy Lifestyles for African Caribbean Women: Reducing Obesity Risks. The one on one interactive session will discuss the association between breast cancer and obesity as well as other major health problems associated with obesity. They learn how to assess their Body Mass Index and measure waist conference to determine whether or not they are at risk for obesity related health problems. The session will last approximately one hour. They will also be briefly reassessed for abuse to determine if abuse is escalating and the need for a referral. Participant contact information will be confirmed and Session 3 scheduled two weeks later.

Session 3: At time three participants in the comparison control health promotion group control will engage in a follow up group session of 6-8 women that will include sharing progress made on developing breast health plans as well as planned choices to reduce obesity and promote healthy lifestyles including diet and exercise. The group discussion will be facilitated by the original facilitator as well as one of the study investigators. Contact information for the final follow up will be will be validated. Participants will complete a post interview on the computer and a 3 month follow-up outcome assessment will be scheduled.

C. Outcome Measures Time 4: Intervention outcomes will be measured at three months to assess effectiveness and safety of the Integrated Risk Reduction Intervention for Women Experiencing IPA. Participants will include women who completed all three sessions of the Risk Reduction intervention or three sessions of the Health Education Comparison Control group. The outcome measures will be completed on computer tablets and will include the same measures that were used at the initial assessment in addition to an assessment of changes in safety and prevention behaviors. Participants will be scheduled for a six month follow-up for final outcome measures.

Time 5: Final post intervention outcome measures will be obtained six months after the participant completes the 3 month outcome measures. The women will again be contacted at least two weeks prior to the scheduled outcomes measures by Caribbean Exploratory NIMHD Research Center Staff to re-confirm the scheduled follow-up and will repeat the same process on computer tablets including outcome measures used at the three month assessment.

D. Data management

1. Preliminary Analyses: Microsoft Access and Excel will be used for record keeping, tracking, and initial data processing. The latest versions of SAS and SPSS computer programs will be used for data management and analysis. Access to the computers and data CDs will be limited both physically and electronically. Computers and data will be stored in an office that is locked when not in use. Access to databases will be restricted with read and write protection. Data analysis will begin with preparatory activities such as the treatment of missing data, identification of outliers and other such data cleaning tasks. A detailed descriptive analysis of all quantitative data will be performed, involving the summarization of data and the use of inferential and graphical exploratory data analytic techniques.
2. Analysis: To conduct a preliminary test of the integrated intervention as described in the brief description, analysis of covariance, frequency and logistic regression will be used to explore potential differences in predictor variables between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Woman: African American/ African Caribbean/African heritage/Mixed
* Age 18 - 44 (A.1)
* Abused (physical, sexual emotional abuse) by an intimate male partner based on responses to screening questions
* Has had an intimate male partner in the last 2 years
* Resident of the US Virgin Islands and plans to remain for next two years

Exclusion Criteria:

* Woman: Not African American/African Caribbean or African Heritage/Mixed
* Under or over age limit
* No intimate partner in the last two years
* No history of physical, sexual or emotional abuse by an intimate partner
* Non resident of US Virgin Islands

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Danger Assessment Score | Change in danger assessment score at three months and six months with significant downward trend
  Danger Assessment (DA-2) The DA-2 is a 20-item scale that assesses the danger of intimate partner homicide for battered women. Danger assessment scores will decrease Internal consistency reliability has ranged between 0.60 to 0.86, with test-retest reliability of 0.89 to 0.94). All research samples have included a substantial portion of minority women (primarily African-American) and women from a variety of clinical and community settings.

SECONDARY OUTCOMES:
Condom Influence Strategies Index | Three months and six month outcome results
  Abused women report increased use of safe sexual behaviors including increased scores on the condom use negotiation scale and increased self-reported practice of sexual safety behaviors..

OTHER OUTCOMES:
Number of participants with Adverse Events Reports as a measure of safety and efficacy | Three months and six months
  Change (decrease) in number of participants reporting incidents physical, sexual and/ or emotional problems related to IPV or IPV and increased use of safety plans and community resources by abused women
Reported sexually transmitted infections and HIV/AIDS | 3 months and six months
  Change (decrease ) in number of abused women reporting an STI's and increased reports of behaviors that reduce risk for HIV among abused women in the integrated risk reduction intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Doris W Campbell, PhD, RN, Principal Investigator — University of the Virgin Islands, Caribbean Exploratory Research Center
Locations (1):
- Caribbean Exploratory NIMHD Research Center,University of the Virgin Islands, School of Nursing, Charlotte Amalie, Virgin Islands

REFERENCES:
- [Background] Campbell J, Jones AS, Dienemann J, Kub J, Schollenberger J, O'Campo P, Gielen AC, Wynne C. Intimate partner violence and physical health consequences. Arch Intern Med. 2002 May 27;162(10):1157-63. doi: 10.1001/archinte.162.10.1157. PMID 12020187
- [Background] Campbell DW, Sharps PW, Gary FA, Campbell JC, Lopez LM. Intimate partner violence in African American women. Online J Issues Nurs. 2002;7(1):5. PMID 12044219
- [Background] Campbell JC, Baty ML, Ghandour RM, Stockman JK, Francisco L, Wagman J. The intersection of intimate partner violence against women and HIV/AIDS: a review. Int J Inj Contr Saf Promot. 2008 Dec;15(4):221-31. doi: 10.1080/17457300802423224. PMID 19051085
- [Background] Jones AS, Dienemann J, Schollenberger J, Kub J, O'Campo P, Gielen AC, Campbell JC. Long-term costs of intimate partner violence in a sample of female HMO enrollees. Womens Health Issues. 2006 Sep-Oct;16(5):252-61. doi: 10.1016/j.whi.2006.06.007. PMID 17055378
- [Background] Brown DS, Finkelstein EA, Mercy JA. Methods for estimating medical expenditures attributable to intimate partner violence. J Interpers Violence. 2008 Dec;23(12):1747-66. doi: 10.1177/0886260508314338. Epub 2008 Feb 26. PMID 18314507
- [Background] Breiding MJ, Black MC, Ryan GW. Prevalence and risk factors of intimate partner violence in eighteen U.S. states/territories, 2005. Am J Prev Med. 2008 Feb;34(2):112-8. doi: 10.1016/j.amepre.2007.10.001. PMID 18201640
- [Background] Krug EG, Mercy JA, Dahlberg LL, Zwi AB. [World report on violence and health]. Biomedica. 2002 Dec;22 Suppl 2:327-36. Spanish. PMID 12596453
- [Background] Gage AJ, Hutchinson PL. Power, control, and intimate partner sexual violence in Haiti. Arch Sex Behav. 2006 Feb;35(1):11-24. doi: 10.1007/s10508-006-8991-0. PMID 16502150
- [Background] Centers for Disease Control and Prevention (CDC). Trends in HIV/AIDS diagnoses--33 states, 2001-2004. MMWR Morb Mortal Wkly Rep. 2005 Nov 18;54(45):1149-53. PMID 16292247
- [Background] Lucea MB, Stockman JK, Mana-Ay M, Bertrand D, Callwood GB, Coverston CR, Campbell DW, Campbell JC. Factors influencing resource use by African American and African Caribbean women disclosing intimate partner violence. J Interpers Violence. 2013 May;28(8):1617-41. doi: 10.1177/0886260512468326. Epub 2013 Jan 6. PMID 23295377
- [Background] Stockman JK, Lucea MB, Draughon JE, Sabri B, Anderson JC, Bertrand D, Campbell DW, Callwood GB, Campbell JC. Intimate partner violence and HIV risk factors among African-American and African-Caribbean women in clinic-based settings. AIDS Care. 2013;25(4):472-80. doi: 10.1080/09540121.2012.722602. Epub 2012 Sep 25. PMID 23006050
- [Background] Campbell JC, Lucea MB, Stockman JK, Draughon JE. Forced sex and HIV risk in violent relationships. Am J Reprod Immunol. 2013 Feb;69 Suppl 1(0 1):41-4. doi: 10.1111/aji.12026. Epub 2012 Oct 16. PMID 23066950
- [Background] Sabri B, Stockman JK, Bertrand DR, Campbell DW, Callwood GB, Campbell JC. Victimization experiences, substance misuse, and mental health problems in relation to risk for lethality among African American and African Caribbean women. J Interpers Violence. 2013 Nov;28(16):3223-41. doi: 10.1177/0886260513496902. Epub 2013 Aug 7. PMID 23929602
- [Background] Draughon JE, Lucea MB, Campbell JC, Paterno MT, Bertrand DR, Sharps PW, Campbell DW, Stockman JK. Impact of Intimate Partner Forced Sex on HIV Risk Factors in Physically Abused African American and African Caribbean Women. J Immigr Minor Health. 2015 Oct;17(5):1313-21. doi: 10.1007/s10903-014-0112-x. PMID 25248623
- [Background] Stockman JK, Lucea MB, Bolyard R, Bertand D, Callwood GB, Sharps PW, Campbell DW, Campbell JC. Intimate partner violence among African American and African Caribbean women: prevalence, risk factors, and the influence of cultural attitudes. Glob Health Action. 2014 Sep 12;7:24772. doi: 10.3402/gha.v7.24772. eCollection 2014. PMID 25226418